CLINICAL TRIAL: NCT04250272
Title: Serratus Anterior Plane Block vs. Intercostal Nerve Block for Postoperative Analgesic Effect After Video-assisted Thoracoscopic Lobectomy: A Randomized Prospective Study
Brief Title: Serratus Anterior Plane Block Versus Intercostal Nerve Block for Postoperative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-07-008-002
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Analgesia; Postoperative Pain; Lung Cancer
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Anterior Plane Block (Experimental): Serratus Anterior Plane Block was performed just before the start of surgery after anesthetic induction through ultrasound-guidance. 20ml of 0.375% ropivacaine was slowly injected between the fascia of serratus anterior and latissimus dorsi near 5th rib.
  Interventions: Procedure: Thoracoscopic lobectomy
- Intercostal Nerve Block (Active Comparator): Intercostal Nerve Block was performed just before closing the surgical incision while looking directly at the affected intercostal space. 10ml of 0.375% ropivacaine was delivered evenly at anterior and posterior intercostal spaces from the port site.
  Interventions: Procedure: Thoracoscopic lobectomy

INTERVENTIONS:
Procedure: Thoracoscopic lobectomy — Thoracoscopic lobectomy was performed for lung cancer

SUMMARY:
A prospective randomized controlled study was undertaken to compare the postoperative analgesic effect between ultrasound-guided serratus anterior plane block and intercostal nerve block after video-assisted thoracoscopic lobectomy.

DETAILED DESCRIPTION:
Post-thoracotomy pain is one of the most notorious postsurgical pains that one can experience. The pain is known to last for an extensive period of time with significantly high intensity.

In field of thoracic surgery, video-assisted thoracoscopic surgery has been played an important role in alleviating the postoperative pain. In field of anesthesiology, various attempts to alleviate post-thoracotomy pain have been tried along advancement of thoracic surgical techniques. It began with postoperative medication of non-steroid anti-inflammatory drugs, opioids and progressed into implementations such as local analgesia, thoracic epidural block, paravertebral block, intercostal nerve block, interpleural block and serratus anterior plane block.

Many analgesic methods have been applied to alleviate postoperative pain in patients who have undergone thoracoscopic surgeries. However, there are no prospective randomized controlled studies between intercostal nerve block and serratus anterior plane block in video-assisted thoracoscopic lobectomy. The main purpose of this study is to compare and analyze the effects between conventional intercostal nerve block and newly introduced serratus anterior plane block in lung cancer patients who have undergone video-assisted thoracoscopic lobectomy.

This prospective study will discover the efficacy and differences between two methods.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* American Society of Anesthesiologists (ASA) I-III class
* Video-assisted thoracoscopic lobectomy

Exclusion Criteria:

* previous history of allergy to local anesthetics
* psychological disorder
* chronic analgesics or sedatives use
* coagulopathy
* The presence of systemic infection or local infection at injection site
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: numeric rating scale | at postanesthesia care unit (PACU)
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Postoperative pain: numeric rating scale | 3 hours later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Postoperative pain: numeric rating scale | 6 hours later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Postoperative pain: numeric rating scale | 12 hours later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Postoperative pain: numeric rating scale | 24 hours later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)

SECONDARY OUTCOMES:
Number of analgesics consumption | through study completion, an average of 1 yea
  If the participant has additional analgesic requirement postoperatively, ketorolac 30mg will be injected intravenously when numeric rating scale score is measured as 4-5, and fentanyl 50# is injected when numeric rating scale score is over 6.
Amount of analgesics consumption | : through study completion, an average of 1 year
  If the participant has additional analgesic requirement postoperatively, ketorolac 30mg will be injected intravenously when numeric rating scale score is measured as 4-5, and fentanyl 50# is injected when numeric rating scale score is over 6.

CONTACTS AND LOCATIONS:
Overall Officials: Saeyoung Kim, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea